CLINICAL TRIAL: NCT02239302
Title: Obstructed Defaecation: Proctography Versus Ultrasound (TPUS and EVUS) in Symptomatic Patients
Brief Title: Obstructed Defaecation: Proctography Versus Ultrasound in Symptomatic Patients
Acronym: OPUS
Status: Completed | Type: Observational
Sponsor: Croydon University Hospital (Other)
Responsible Party: Principal Investigator, Ranee Thakar, Consultant Urogynaecologist, Croydon University Hospital
Other Study IDs: 13/LO/1665
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Obstructed Defaecation Syndrome
Keywords: Obstructed defaecation syndrome; Transperineal Ultrasound; Endovaginal Ultrasound; Evacuation Proctography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Obstructed defaecation syndrome is a common problem in which patients experience difficulty to evacuate stools and feel that the bowel is incompletely empty, which causes the need to put fingers in to the rectum or vaginal to empty the rectum. These symptoms have a significant effect on social, physical, emotional and sexual wellbeing all of which have impact on quality of life. These symptoms are caused by posterior compartment disorders such as the last part of the large bowel bulging into the vagina (rectocele), the small bowel pressing on the rectum (enterocele), a circumferential infolding of the rectal wall (intussusception) or paradoxical pelvic floor contraction during attempts to evacuate (anismus).

Currently the evacuation proctogram is the gold standard for diagnosis of posterior compartment disorders. This technique, however, exposes the patient to ionising radiation, requires preparation of the small and large bowel with contrast and defaecation in a non-private setting, which most women find embarrassing and unpleasant. Over the years, research has focussed on identifying alternatives that are better tolerated to substitute evacuation proctography. Ultrasound is a widely available, non-expensive, non-invasive, fast and a well-tolerated method for the dynamic and static imaging of the pelvic floor without the use of ionising radiation. The level of agreement between transperineal ultrasound (TPUS) and proctography for varies widely. Endovaginal ultrasound (EVUS) not yet compared to proctography. The aim of this study is to assess the level of agreement between ultrasound (EVUS and TPUS) and evacuation proctography in the diagnosis of posterior compartment disorders.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Symptoms of obstructed defaecation
* Planned for evacuation proctography

Exclusion Criteria:

* Inability to understand English
* Unwilling to consent for evacuation proctography
* Under 18 years of age
* Virgo intacta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with symptomes of obstructed defaecation
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the level of agreement between ultrasound (EVUS and TPUS) and evacuation proctography in the diagnosis of posterior compartment disorders | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ranee Thakar, FRCOG, Principal Investigator — Croydon University Hospital
Locations (1):
- Croydon University Hospital, Croydon, Surrey, United Kingdom

REFERENCES:
- [Derived] van Gruting IMA, Stankiewicz A, Kluivers K, De Bin R, Blake H, Sultan AH, Thakar R. Accuracy of Four Imaging Techniques for Diagnosis of Posterior Pelvic Floor Disorders. Obstet Gynecol. 2017 Nov;130(5):1017-1024. doi: 10.1097/AOG.0000000000002245. PMID 29016504